CLINICAL TRIAL: NCT06560346
Title: Understanding the Natural History Early in the Course or Presentation of Friedreich Ataxia (EARLY-FA); Evaluating New Clinical Outcome Assessments in Children With Friedreich Ataxia to Facilitate Clinical Trial Design.
Brief Title: Understanding the Natural History Early in the Course or Presentation of Friedreich Ataxia
Acronym: EARLY-FA
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funding
Sponsor: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-025
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Friedreich Ataxia; Rare Diseases
MeSH Terms: conditions — Friedreich Ataxia; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Whole blood and plasma will be collected to assess frataxin and lipids in FRDA patients and controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FRDA, genetically confirmed: individuals with FRDA, genetically confirmed, aged 4-21yrs
  Interventions: Other: Geneticlly confirmed disease causing FXN mutatuion
- Matched healthy controls: Participants in the control group (Group 2) will be aged 4-21 years at enrollment and fulfill group matching criteria to an enrolled participant with FRDA (age, sex)
  Interventions: Other: Healthy Control

INTERVENTIONS:
Other: Geneticlly confirmed disease causing FXN mutatuion — No intervention in this observational Natural History Study
  Groups: FRDA, genetically confirmed
Other: Healthy Control — No intervention in this observational Natural History Study
  Groups: Matched healthy controls

SUMMARY:
Multicenter, prospective, observational natural history and outcome measure study of children and young adults with Friedreich ataxia.

DETAILED DESCRIPTION:
A multicenter, prospective, observational natural history and outcome measure study of children and young adults with Friedreich ataxia to further understand the disease features and progression and inform and enable future clinical trials in children with FA.

The study, Understanding the natural history early in the presentation of Friedreich ataxia: evaluating new clinical outcome assessments in children with Friedreich ataxia to facilitate clinical trial design (EARLY-FA), evaluates disease features specific to children and novel biomarkers and outcome measures which leveraging existing clinical research infrastructure and data collection from an established natural history study, UNIFAI.

ELIGIBILITY:
Inclusion criteria for participants with FA:

1. Genetic diagnosis of Friedreich Ataxia
2. Ages 4-21 years at enrollment
3. Enrollment in the UNIFAI study and ability to have simultaneous visits for both UNIFAI and EARLY-FA
4. Informed consent must be obtained for all participants:

   1. For underage participants, they and the parent/ legally authorized representative have to sign the informed consent form, child assent (if applicable)
   2. Persons who are not legally competent require the informed consent of their legally authorized representative

Inclusion criteria for control participants:

1. Ages 4-21 years at enrollment
2. Matching criteria to an enrolled participant with FA (age, sex and educational status)
3. Informed consent must be obtained for all participants:

   1. For underage participants, they and the parent/ legally authorized representative have to sign the informed consent form, child assent (if applicable)
   2. Persons who are not legally competent require the informed consent of their legally authorized representative

Exclusion criteria for participants with FA:

1. Diagnosis of non-FA medical or other condition that in the opinion of the investigator would interfere with the conduct and assessments of the study or be confounding and contraindication to participation.
2. Pregnant female participants
3. Unable to provide informed consent.

Exclusion criteria for control participants:

1. Family risk for FA with unknown status
2. Diagnosis of a medical condition that in the opinion of the investigator could be confounding and contraindication to participation
3. Unable to provide informed consent

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will enroll 200 individuals with FA who are 4-21 years of age and 100 healthy matched (age and sex) controls.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between growth (height in z-score) and disease severity in FRDA (mFARS score) | Baseline, 12 months, and 24 months
  Height (cm) will be measured using a wall-mounted stadiometer and univariate analyses will test for Correlation between the height Z-score (after accounting for genetic potential (mid-parental height)) and disease severity (using the standard ataxia scale modified Friedreichs ataxia rating scale (mFARS)).
  The modified Friedreich Ataxia Rating Scale (mFARS) is a disease-specific scale that measures progression of neurological effects of FA. The mFARS is a validated and reliable scale; comprised of the neurologic component of the FARS and evaluates bulbar, upper limb, lower limb, and upright stability/gait function. For each item, responses categorize the corresponding neurological finding, and the findings are assigned a score ranging from 0 to 3, 4, or 5 with 0 being normal and higher numbers indicative of greater impairment. The score ranges from 0 to 93. The score will be compared to the previous year annually for up to 25 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Farmer, Study Director — Friedreich's Ataxia Research Alliance
Locations (7):
- United States (3):
  - University of Iowa, Stead Family Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia
- McGill University Health Centre - Montreal Neurological Institute, Montreal, Quebec, Canada
- University Hospital Aachen, Dept. of Neurology, Aachen, Germany
- Bambino Gesù Children's Hospital, Department of Neurosciences, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
All such study data will be made available to all study investigators after it has been generated, per the policies outlined in the study agreements and for analysis. The sponsor plans to make de-identified data available to third parties at the conclusion of the study and after primary manuscripts have been published, including depositing data in a secure platform.
  All de-identified dataset(s) that can be shared will be deposited in the Rare Disease Cures Accelerator Data and Analytics Platform (RDCA-DAP) hosted and managed by the Critical Path Institute (C-Path). RDCA-DAP is an FDA-funded initiative that provides a centralized and standardized infrastructure to support and accelerate rare disease characterization with the goal of accelerating therapy development.
  Each site will be required to ensure that participants are consented in such a way that allows the sharing of de-identified data with the community in this manner.
Supporting Information: Study Protocol
Time Frame: At the conclusion of the study and after primary manuscripts have been published
Access Criteria: Access and requests managed by the RDCA DAP platform